CLINICAL TRIAL: NCT03093155
Title: A Randomized Phase II Evaluation of Weekly Ixabepilone With or Without Biweekly Bevacizumab in Recurrent or Persistent Platinum-resistant/Refractory Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancers
Brief Title: Evaluation of Weekly Ixabepilone With or Without Biweekly Bevacizumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: R-Pharm US LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000020232
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — ixabepilone; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ixabepilone (Active Comparator): Ixabepilone 20 mg/m2 days 1, 8, 15 Q 28 days
  Interventions: Drug: Ixabepilone
- Ixabepilone + Bevacizumab (Experimental): Ixabepilone 20 mg/m2 days 1, 8, 15
  + Bevacizumab 10 mg/kg days 1, 15 Q 28 days
  Interventions: Drug: Ixabepilone; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ixabepilone — Ixabepilone will be administered at 20 mg/m2 intravenously days 1, 8, 15 of a 28-day cycle over one hour.
  Treatment will continue until progression, death, or prohibitive side effects. If any patient has a complete response, patient may stop treatment after 2 additional consolidation cycles following documented complete response
  Other Names: Ixempra
Drug: Bevacizumab — Bevacizumab will be administered at 10 mg/kg intravenously days 1, 15 of a 28-day cycle over one hour. Bevacizumab will be infused after ixabepilone. The first dose of bevacizumab will be administered intravenously over 90 minutes; the second dose may be administered over 60 minutes if no prior reaction to previous infusion; subsequent doses may be administered over 30 minutes if no prior reaction to previous infusion.
  Treatment will continue until progression, death, or prohibitive side effects. If any patient has a complete response, patient may stop treatment after 2 additional consolidation cycles following documented complete response.
  Other Names: Avastin
  Arms: Ixabepilone + Bevacizumab

SUMMARY:
This is a randomized, two-arm, open-label Phase II multicenter study designed to examine the effects of adding bevacizumab to ixabepilone for the treatment of patients who have recurrent or persistent platinum-resistant/refractory epithelial (non-mucinous) ovarian, fallopian tube, or primary peritoneal cancer. Its primary objective is to assess whether adding bevacizumab to ixabepilone improves progression-free survival in its target population. Study participants will be stratified by (a) study site and (b) previous receipt of bevacizumab prior to randomization.

DETAILED DESCRIPTION:
The primary objective of this study is as follows:

* To assess the activity of ixabepilone with bevacizumab compared to ixabepilone alone in patients with recurrent or persistent platinum-resistant/refractory epithelial (non-mucinous) ovarian, fallopian tube, or primary peritoneal cancer. We will assess this by comparing the ixabepilone +bevacizumab (experimental) arm to the ixabepilone-alone (control) arm for an improvement in median progression free survival (PFS).

The secondary objectives of this study are as follows:

* To compare the experimental arm to the control arm for increases in objective response rate (ORR) and durable disease control rate (DDCR).
* To compare the experimental arm to the control arm for an increase in overall survival (OS).
* To assess the safety profile of ixabepilone in combination with bevacizumab in ovarian, fallopian tube, or primary peritoneal cancer patients.
* To assess whether prior treatment with bevacizumab impacts future response to bevacizumab in combination with ixabepilone.

In addition to the primary and secondary objectives of this study, there are additional exploratory/correlative objectives. The exploratory/correlative objectives of this study are as follows:

* To characterize number, length and composition (e.g., class III β-tubulin expression) of microtentacles (McTNs) isolated from circulating tumor cells isolated from whole blood of patients undergoing treatment with ixabepilone with or without bevacizumab, and correlate with best response, PFS, and OS.
* To observe McTNs on circulating tumor cells in blood using a novel polyelectrolyte multi-layer (PEM) tethering technology.
* To correlate ex vivo response of McTNs to drug treatment with clinical response in order to develop a real-time assay to predict response to therapy.
* To explore use of circulating tumor (ct) DNA as a biomarker for disease response and compare its performance to CA-125.
* To examine whether clinical response to ixabepilone with or without bevacizumab differs between high and low expressors of class III β-tubulin.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have platinum-resistant/refractory (i.e., platinum-free interval <6 months) recurrent or persistent histologically confirmed epithelial (non-mucinous) ovarian, fallopian tube, or primary peritoneal cancer.

Patients may have serous, endometrioid, clear cell, carcinosarcoma, or transitional cell/malignant Brenner, mixed, or undifferentiated histologies.

* Patients must have specimen available for immunohistochemistry for class III β-tubulin status; recurrent tumor specimen is preferred, though this may be performed on primary tumor if no recurrent tumor is available.
* All patients must have measurable disease. Measurable disease is defined as lesions that can be measured by physical examination or by means of medical imaging techniques. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation or plain x-ray, or ≥ 10 mm when measured by spiral CT and/or MRI. Ascites and pleural effusions are not to be considered measurable disease.
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST v1.1 Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* At the time of initial surgery, patients may have been optimally (<1 cm diameter residual disease) or sub-optimally (≥1 cm diameter of residual disease) debulked.
* Patients with measurable recurrent disease of any previous stage (I-IV) are eligible to enrollment.
* The diagnosis must be histologically confirmed by a gynecologic pathologist.
* Patients must have adequate bone marrow, kidney, and liver function:

  1. Absolute neutrophil count greater than or equal to 1500 cells/mm3
  2. Platelets greater than or equal to 100,000/uL
  3. Renal function: creatinine less than or equal to 2.0 mg/dL
  4. Hepatic function: Bilirubin ≤ 1.5 X laboratory normal
  5. SGOT/SGPT ≤ 3 X laboratory normal.
* Patients must have an ECOG performance status of 0-2.
* Patients must have signed an approved informed consent.
* Patients must have recovered from effects of recent surgery, radiotherapy, or chemotherapy. They should be free of significant infection.
* Patients must have received prior treatment with taxanes. There is no limit on the number of prior lines of therapy.
* Patients may have received prior bevacizumab therapy alone or in combination with chemotherapy. A 3-week washout period is required.
* Patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to the study entry and be practicing an effective form of contraception (section 7.5.3).
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancers, are excluded if there is any evidence of other malignancy present within the last five years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Patients who have a significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure, or uncontrolled arrhythmias within 6 months of registration (NYHA classification III-IV).
* Patients with any unstable medical issue (including cardiac issues as above, active treatment for symptomatic pulmonary embolism, CVA, renal or hepatic insufficiency, active infection/sepsis requiring intravenous antibiotics). In patients who have undergone surgery, 28 days should elapse before initiation and the surgical site should be adequately healed.
* Known brain/leptomeningeal involvement of the disease, active neurological disease such as uncontrolled seizure disorder or moderate to severe dementia.
* Patients who have received prior therapy with any covalent irreversible anti-angiogenic tyrosine kinase inhibitor (e.g., vandetanib).
* Patients known to be seropositive for human immunodeficiency virus (HIV) and active hepatitis, even if liver function studies are in the eligible range.
* Known hemorrhagic diathesis or active bleeding disorder, including platelet count <100,000/uL, or inadequate granulocytes, including an absolute neutrophil count <1500 cells/mm.
* Any hypersensitivity to Cremophor® EL or polyoxyethylated castor oil.
* CTCAE grade 2 or higher peripheral neuropathy.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 78 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D. Santin, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Marlene & Stewart Greenebaum Comprehensive Cancer Center, University of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Roque DM, Siegel ER, Buza N, Bellone S, Silasi DA, Huang GS, Andikyan V, Clark M, Azodi M, Schwartz PE, Rao GG, Reader JC, Hui P, Tymon-Rosario JR, Harold J, Mauricio D, Zeybek B, Menderes G, Altwerger G, Ratner E, Santin AD. Randomised phase II trial of weekly ixabepilone +/- biweekly bevacizumab for platinum-resistant or refractory ovarian/fallopian tube/primary peritoneal cancer. Br J Cancer. 2022 Jun;126(12):1695-1703. doi: 10.1038/s41416-022-01717-6. Epub 2022 Feb 11. PMID 35149854
- [Derived] Roque DM, Siegel ER, Buza N, Bellone S, Huang GS, Altwerger G, Andikyan V, Clark M, Azodi M, Schwartz PE, Rao GG, Ratner E, Santin AD. Randomized phase II trial of weekly ixabepilone +/- biweekly bevacizumab for platinum-resistant or refractory ovarian/fallopian tube/primary peritoneal cancer (NCT03093155): Updated survival and subgroup analyses. BJC Rep. 2024 Jun 20;2(1):43. doi: 10.1038/s44276-024-00067-5. PMID 39516558
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone: Ixabepilone 20 mg/m2 days 1, 8, 15 Q 28 days
  Ixabepilone: Ixabepilone will be administered at 20 mg/m2 intravenously days 1, 8, 15 of a 28-day cycle over one hour.
  Treatment will continue until progression, death, or prohibitive side effects. If any patient has a complete response, patient may stop treatment after 2 additional consolidation cycles following documented complete response
- Ixabepilone + Bevacizumab: Ixabepilone 20 mg/m2 days 1, 8, 15
  + Bevacizumab 10 mg/kg days 1, 15 Q 28 days
  Ixabepilone: Ixabepilone will be administered at 20 mg/m2 intravenously days 1, 8, 15 of a 28-day cycle over one hour.
  Treatment will continue until progression, death, or prohibitive side effects. If any patient has a complete response, patient may stop treatment after 2 additional consolidation cycles following documented complete response
  Bevacizumab: Bevacizumab will be administered at 10 mg/kg intravenously days 1, 15 of a 28-day cycle over one hour. Bevacizumab will be infused after ixabepilone. The first dose of bevacizumab will be administered intravenously over 90 minutes; the second dose may be administered over 60 minutes if no prior reaction to previous infusion; subsequent doses may be administered over 30 minutes if no prior reaction to previous infusion.
  Treatment will continue until progression, death, or prohibitive side effects. If any patient has a complete response, patient may stop treatment after 2 additional consolidation cycles following documented complete response.
Period: Overall Study
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Started | 38 | 40
Patients Completing Treatment | 37 | 39
Patients Requiring Dose Reduction | 21 | 25
Completed | 37 | 39
Not Completed | 1 | 1
Not completed — Not Eligible | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only those that remained on study are included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Continuous [Median (Full Range); unit: years] | 67 [50 to 88] | 67 [40 to 78] | 67 [40 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 39 | 76
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 34 | 37 | 71
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 27 | 31 | 58
  Race: Black | 8 | 4 | 12
  Race: Other | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 37 | 39 | 76
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group Performance Status (ECOG PS) scale ranges from 0 to 5. 0: Fully active; 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work; 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4: Completely disabled. Cannot carry out any self-care. Totally confined to bed or chair; 5: Dead.
  Participants
    0-1 | 31 | 36 | 67
    2 | 6 | 3 | 9
Histology [Count of Participants; unit: Participants]
  Serous | 29 | 34 | 63
  Carcinosarcoma | 2 | 1 | 3
  Other | 6 | 4 | 10
Prior Lines of Chemotherapy [Count of Participants; unit: Participants]
  Less than or Equal to 3 | 18 | 21 | 39
  Greater than 3 | 19 | 18 | 37
Prior Bevacizumab [Count of Participants; unit: Participants]
  Yes | 21 | 21 | 42
  No | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Differences Between Ixabepilone Alone and Ixabepilone + Bevacizumab
Description: Progression-free survival (PFS), the primary endpoint, will be defined as the length of time from randomization to disease recurrence, disease progression, or death for any reason. The timeframe was updated upon results entry.
Time Frame: Up to 37 months
Population: Those completing treatment post randomization
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Number analyzed (Participants) | 37 | 39
months | 2.20 [1.61 to 4.96] | 5.46 [3.98 to 11.47]
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Bevacizumab; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.31, 90% CI 2-sided [0.20 to 0.49]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Treatment response will be based on RECIST v1.1 Guidelines for measurable lesions. Objective response rate (ORR) includes evaluation for partial response (PR) or complete response (CR). Time frame was updated upon results entry.
Time Frame: Up to 37 months
Population: Those completing treatment post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Number analyzed (Participants) | 37 | 39
Participants | 3 | 15
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Bevacizumab; Test type: Superiority; p = 0.003, Fisher Exact

3. Secondary Outcome: Overall Survival (OS) Differences Between Ixabepilone Alone and Ixabepilone + Bevacizumab
Description: Overall survival (OS) is defined as time from randomization to death from any cause. Time frame was updated upon results entry.
Time Frame: Up to 37 months
Population: Those completing treatment post randomization
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Number analyzed (Participants) | 37 | 39
months | 6.05 [2.83 to 16.80] | 10.32 [7.92 to 28.14]
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Bevacizumab; Test type: Superiority; p = 0.018, Regression, Cox; Hazard Ratio (HR) = 0.56, 90% CI 2-sided [0.38 to 0.84]

4. Secondary Outcome: Number of Participants With Treatment Related SAEs
Description: Safety profile of Ixabepilone in combination with Bevacizumab as defined by Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Presented are the number of participants that experienced SAE's related to study drug. Full reporting of adverse events is presented in the Adverse Events module. Time frame was updated upon results entry.
Time Frame: Up to 37 months
Population: Those completing treatment post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Number analyzed (Participants) | 37 | 39
Participants | 6 | 8
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Bevacizumab; Test type: Superiority; p = 0.77, Fisher Exact

5. Secondary Outcome: Differences in Response to the Combination of Ixabepilone and Bevacizumab in Relationship to Previous Treatment With Bevacizumab and Taxanes
Description: Assess whether prior treatment with Taxanes impacts future response to Bevacizumab in combination with Ixabepilone. BEST RESPONSE using RECIST Criteria- Complete Response (CR): The disappearance of all target lesions. There should be no evidence of disease, and any pathological lymph nodes must have reduced in size to normal (short axis less than 10 mm). Partial Response (PR): At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since the treatment started. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesion
Time Frame: Up to 41 months
Population: Those with prior Taxanes treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Number analyzed (Participants) | 13 | 10
Participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 3
  Stable Disease (SD) | 7 | 6
  Progressive Disease (PD) | 5 | 1
  Not Assessed | 1 | 0
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Bevacizumab; The RECIST responses were categorized as SD/PD or NA compared to PR or Better as a binary outcome; Test type: Superiority; p = 0.068, Fisher Exact

6. Secondary Outcome: Durable Disease Control Rate (DDCR) Differences Between Ixabepilone Alone and Ixabepilone + Bevacizumab
Description: Treatment response will be based on RECIST v1.1 Guidelines for measurable lesions. Objective response rate (ORR) includes evaluation for partial response (PR) or complete response (CR).
  Durable Disease Control (DDC) is defined as complete response (CR), partial response (PR), or stable disease (SD) ≥6 months from date of best response. Presented are the counts of those that achieved DDC.
Time Frame: 5 Years
Population: Those completing treatment post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
Number analyzed (Participants) | 37 | 39
Participants | 1 | 14

ADVERSE EVENTS:
Time Frame: Up to 37 months
Arm/Group | Ixabepilone | Ixabepilone + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 36/37 | 34/39
Serious Adverse Events (participants affected / at risk) | 24/37 | 16/39
Other Adverse Events (participants affected / at risk) | 36/37 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone (N=37) | Ixabepilone + Bevacizumab (N=39)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 5 (5) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixabepilone (N=37) | Ixabepilone + Bevacizumab (N=39)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5 (5) | 10 (21)
Anemia (Blood and lymphatic system disorders) | 6 (8) | 8 (15)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 4 (4)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (5)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 25 (38) | 30 (41)
Diarrhea (Gastrointestinal disorders) | 22 (36) | 23 (40)
Vomiting (Gastrointestinal disorders) | 20 (28) | 17 (27)
Constipation (Gastrointestinal disorders) | 9 (9) | 17 (19)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 15 (20)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7 (7) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 9 (10) | 4 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (2) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 24 (53) | 36 (79)
General disorders and administration site conditions - Other, specify (General disorders) | 12 (14) | 11 (11)
Edema limbs (General disorders) | 8 (9) | 5 (5)
Pain (General disorders) | 4 (4) | 7 (7)
Infusion related reaction (General disorders) | 2 (2) | 3 (7)
Fever (General disorders) | 2 (3) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (15) | 9 (10)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 5 (5)
Lung infection (Infections and infestations) | 4 (4) | 3 (4)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Skin infection (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory infection (Infections and infestations) | 0 (0) | 4 (4)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (4) | 3 (3)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 10 (13)
Creatinine increased (Investigations) | 4 (6) | 6 (6)
Neutrophil count decreased (Investigations) | 3 (5) | 6 (12)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 17 (17) | 20 (25)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (15) | 9 (15)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 3 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 10 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (10) | 25 (32)
Headache (Nervous system disorders) | 2 (2) | 11 (13)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 4 (6)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 5 (5) | 6 (6)
Proteinuria (Renal and urinary disorders) | 0 (0) | 8 (16)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (3) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 13 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 17 (25)
Hypotension (Vascular disorders) | 1 (1) | 5 (6)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03093155/Prot_SAP_000.pdf